CLINICAL TRIAL: NCT01173562
Title: An Open-Label, Single-Dose Study to Assess the Safety of 500-mg Mebendazole Chewable Formulation in Children 2 to 10 Years of Age, Inclusive
Brief Title: A Safety Study of Mebendazole in Children 2 to 10 Years of Age
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR017419; MEBENDAZOLGAI3002 (Other: Johnson & Johnson Pharmaceutical Research & Development, L.L.C.)
Record Dates: First submitted 2010-07-29; First posted 2010-08-02 (Estimated); Last update posted 2014-03-12 (Estimated); Status verified 2014-03

CONDITIONS: Healthy Volunteers
Keywords: Healthy volunteers; Parasitic Diseases; Mebendazole (VERMOX); Anthelmintics; Antiparasitic Agents; Soil-transmitted helminth (STH) infections; Pediatric
MeSH Terms: conditions — Parasitic Diseases; Infections | interventions — Mebendazole

ARMS (1):
- Mebendazole (Experimental)
  Interventions: Drug: Mebendazole

INTERVENTIONS:
Drug: Mebendazole — Type= exact number, unit= mg, number= 500, form= chewable tablet, route= oral use. One mebendazole 500-mg chewable tablet taken on Day 1.

SUMMARY:
The purpose of this study is to assess the safety and tolerability of mebendazole 500-mg chewable tablet formulation in a pediatric population. Mebendazole is a drug used for the treatment of soil-transmitted parasitic helminth (STH) (ie, parasitic worm) infections such as pinworm, whipworm, common roundworm, common hookworm, and American hookworm.

DETAILED DESCRIPTION:
This is an open-label (identity of study drug will be known to study participant and investigator), single-center, single-dose, single-arm (ie, 1 treatment group) safety study. This study will consist of a screening visit on Day 1 at which time all study-related screening procedures will be performed. After all results are reviewed, children who meet all of the inclusion criteria and none of the exclusion criteria will be entered into the open-label phase of the study. A single mebendazole 500-mg chewable tablet will be administered on Day 1 and the children will remain at the study site so that adverse events can be recorded at approximately 30 minutes postdose. Study participants will return to the study site 3 days (plus or minus 1 day) postdose at which time adverse events will be recorded again. Safety will be monitored during the study by assessing adverse events by direct observation at 30 minutes after dosing and at 3 days (plus or minus 1 day) after dosing, by direct observation of the study participant, report by the parent or guardian, or both. On Day 1, a single mebendazole 500-mg chewable tablet will be chewed and swallowed by each study participant. If desired, study participants will be allowed to drink water when administered study drug.

ELIGIBILITY:
Inclusion Criteria:

* Be an otherwise healthy child based on medical history, physical examination, vital signs, and concomitant medications and live in a high-prevalence area where parasite infection is endemic (ie, Prevalent in or peculiar to a particular locality, region, or people)
* Have teeth and be able to chew the mebendazole chewable tablet
* Girls must be premenarchal
* Parent(s)/guardians of study participants (or their legally-accepted representatives) must have signed an informed consent document indicating that they understand the purpose of and procedures required for the study and are willing to have their child participate in the study

Exclusion Criteria:

* Have a history of clinically significant liver or renal insufficiency
* cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurologic, hematologic (eg, anemia), rheumatologic, psychiatric, or metabolic disturbances that, in the opinion of the investigator, renders the candidate not suitable for mebendazole treatment
* Have a suspected massive intestinal parasitic infection, based on history and physical findings, as determined by the principal investigator
* Have any condition that, in the opinion of the investigator, would compromise the well-being of the study participant or the study or prevent the study participant from meeting or performing study requirements

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 397 (Actual)
Dates: Start 2010-02; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
The number, severity, relationship to study drug, and type of adverse events reported. | Baseline (Day 1) to the end of study (Day 3) or early withdrawal visit

SECONDARY OUTCOMES:
Change in physical examination | Baseline (Day 1) to the end of study (Day 3) or early withdrawal visit
Change in vital sign measurements | Baseline (Day 1) to the end of study (Day 3) or early withdrawal visit

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (1):
- Pemba, Tanzania

REFERENCES:
- See also: A Safety Study of Mebendazole in Children 2 to 10 Years of Age — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=863&filename=CR017419_CSR.pdf